CLINICAL TRIAL: NCT05916547
Title: Safety and Efficacy of Extracorporeal Shock Wave Lithotripsy and Endoscopic Retrograde Cholangiopancreatography for Pancreatic Stones
Brief Title: Safety and Efficacy of P-ESWL and ERCP
Status: Completed | Type: Observational
Sponsor: Changhai Hospital (Other)
Responsible Party: Principal Investigator, Zhaoshen Li, Professor, Changhai Hospital
Other Study IDs: SEEPS
Record Dates: First submitted 2023-06-15; First posted 2023-06-23 (Actual); Last update posted 2024-07-11 (Actual); Status verified 2024-07

CONDITIONS: Pancreatic Duct Stone
Keywords: Pancreatic Duct Stone; Pancreatic extracorporeal shock wave lithotripsy; Safety; Efficacy; endoscopic retrograde cholangiopancreatography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: pancreatic extracorporeal shock wave lithotripsy — Pancreatic extracorporeal shock wave lithotripsy is based on the principle of shock wave energy. Whenever energy is abruptly released in an enclosed space, shock waves are generated and then cross to the surface of pancreatic duct stones to cause further fragmentation.

SUMMARY:
To determine the types, incidence and risk factors of adverse events after pancreatic extracorporeal shock wave lithotripsy (P-ESWL) and endoscopic retrograde cholangiopancreatography (ERCP), define the grading criteria of adverse events after P-ESWL and ERCP, and analyze the efficacy of P-ESWL and ERCP, which will provide evidence-based medical evidence to guide physicians' clinical practice.

DETAILED DESCRIPTION:
Currently, pancreatic extracorporeal shock wave lithotripsy (P-ESWL) and endoscopic retrograde cholangiopancreatography (ERCP) has become the preferred treatment for pancreatic duct stones. Although some studies had confirmed the safety and efficacy of P-ESWL and ERCP, the sample size were small and the follow-up period were short. Therefore, investigators designed this study with a large sample and a long follow-up period to clarify the efficacy and safety of P-ESWL and ERCP, so as to guide clinical work, standardize the diagnosis and treatment process of adverse events.

ELIGIBILITY:
Inclusion Criteria:

* Patients hospitalized in Changhai Hospital from 2011.03.01 to 2018.06.30.
* Painful patients with chronic pancreatitis.
* Patients who completed pancreatic extracorporeal shock wave lithotripsy.

Exclusion Criteria:

* Patients who diagnosed pancreatic cancer within 2 years after diagnosing chronic pancreatitis.
* Patients who refused to participate in the study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients hospitalized in Changhai Hospital from 2011.02.01 to 2018.06.30.
Sampling Method: Non-Probability Sample
Enrollment: 2071 (Actual)
Dates: Start 2023-06-01 (Actual); Primary Completion 2024-04-26 (Actual); Study Completion 2024-05-01 (Actual)

PRIMARY OUTCOMES:
the incidence of post-ESWL adverse events | 1 months
  An adverse event of P-ESWL is classified as either a complication or a transient adverse event (TAE), depending on severity. Complications are recognized as adverse events needing specific medical intervention and prolonged hospitalization, while TAEs are defined as transient injuries caused by shock waves, which required no medical intervention and do not prolong hospitalization.

SECONDARY OUTCOMES:
the rate of pancreatic duct clearance | 1 week
  Complete clearance: more than 90% clearance of stone volume; partial clearance: 50% to 90% clearance of stone volume; unsuccessful clearance: failure to fragment the stones to less than 3 mm diameter or less than 50% clearance of stone volume.
Pain relief of patients after P-ESWL and ERCP | more than 24 months
  The ratio of patients with complete pain relief (an Izbicki pain score was ≤ 10), partial relief (an Izbicki pain score > 10 with a decrease of > 50%) and no relief.

CONTACTS AND LOCATIONS:
Overall Officials: Liang-hao Hu, MD, Principal Investigator — Changhai Hospital
Locations (1):
- Changhai Hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Li BR, Liao Z, Du TT, Ye B, Zou WB, Chen H, Ji JT, Zheng ZH, Hao JF, Jiang YY, Hu LH, Li ZS. Risk factors for complications of pancreatic extracorporeal shock wave lithotripsy. Endoscopy. 2014 Dec;46(12):1092-100. doi: 10.1055/s-0034-1377753. Epub 2014 Sep 24. PMID 25251205
- [Derived] Liu Y, Yi JH, Wang PY, Fu P, Kang Y, Wang T, Zhang D, Zhang XH, Xu JJ, Zhang SL, Han PD, Wang F, Zhou XY, Feng JS, Xu JJ, Qian JH, Wang D, Chen H, Liu RH, Wang FY, Li ZS, Hu LH. Safety evaluation of extracorporeal shockwave lithotripsy for pancreatic stones: Experience based on a large chronic pancreatitis cohort. Dig Liver Dis. 2025 Feb;57(2):417-426. doi: 10.1016/j.dld.2024.08.043. Epub 2024 Sep 11. PMID 39261265
- [Derived] Liu Y, Yin XY, Cui JH, Wang T, Feng XY, Yi JH, Xu JJ, Zhang SL, Han PD, Wang D, Liu RH, Wang FY, Li ZS, Hu LH. Long-term clinical outcomes of extracorporeal shockwave lithotripsy and endoscopic retrograde cholangiopancreatography for pancreatic duct stone treatment in patients with chronic pancreatitis. Aliment Pharmacol Ther. 2024 Oct;60(8):1110-1121. doi: 10.1111/apt.18224. Epub 2024 Aug 21. PMID 39169663